CLINICAL TRIAL: NCT05087069
Title: A Phase I, Single-centre, Double-blind, Randomised, Placebo-controlled Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics of BV100 Administered as Multiple Intravenous Doses to Healthy Male Subjects
Brief Title: Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics of BV100 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioVersys SAS (Industry)
Collaborators: Nuvisan GmbH (Unknown)
Responsible Party: Sponsor
Organization: BioVersys AG (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BV100-02
Record Dates: First submitted 2021-10-09; First posted 2021-10-21 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BV100 (Experimental): BV100 intravenous infusion
  Interventions: Drug: BV100
- Placebo (Placebo Comparator): Saline intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BV100 — Rifabutin for Infusion
  Arms: BV100
Drug: Placebo — Saline intravenous infusion
  Arms: Placebo

SUMMARY:
Safety and tolerability and Pharmacokinetics of multiple doses of BV100 in healthy volunteers

DETAILED DESCRIPTION:
The study will investigate the safety and tolerability of increasing multiple intravenous doses of BV100 by assessing the Incidence of treatment-emergent adverse events (TEAEs). In addition the goal is to characterize the multiple dose pharmacokinetic profiles of rifabutin in plasma.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 to 55 years of age inclusive at the time of signing the informed consent.
2. Subjects who are healthy as determined by the Investigator based on medical evaluation including medical history, physical and neurological examination, vital signs, ECG, and clinical laboratory tests at screening and on Day -1.
3. Subjects are able to have an intravenous line placed.
4. Body weight of at least 50 kg and BMI within the range of 19 to 30 kg/m2 (inclusive) at screening examination.
5. Male subjects will be included in the trial.
6. Subjects must agree to the following from the time of the first dose until 3 months after the follow-up visit:

   * use two acceptable methods of birth control with a female partner of child bearing potential (barrier method combined with an additional highly effective contraceptive method). Barrier methods of contraception include condom or occlusive cap (diaphragm or cervical/vault caps). Highly effective contraception is defined in accordance with the Clinical Trial Facilitation Group (CTFG 2020 ) guidance and includes the following methods: hormonal implants, injectables, hormonal intrauterine device, combined hormonal contraceptives, sexual abstinence and vasectomised sexual partner. For details refer to Appendix 2.
   * refrain from donating sperm.
7. Prior to any clinical trial specific procedure the subject provided written informed consent. Subjects must be able to read, write, and fully understand the German language.
8. The subject is a non-smoker, former smoker (<10 pack year smoking history) or former user of nicotine containing products or stable non-smoker for at least 3 months before the first study drug administration. Subjects should also have abstained from use of e-cigarettes for at least 3 months before first study drug administration.

Exclusion Criteria:

1. History of clinically relevant disease of any organ system that may interfere with the objectives of the trial or provide a risk to the health of the subject.
2. Known or suspected history of hypersensitivity to rifabutin or excipients or to drugs of a similar chemical class including rifampicin, rifapentine, rifaximin; history of allergic reactions leading to hospitalisation or any other allergic conditions (including drug allergies, asthma, eczema, anaphylactic reactions but excluding untreated, asymptomatic, seasonal allergies) which the Investigator considers may affect the safety of the subject and/or outcome of the trial.
3. History of antibiotic associated diarrhoea within the last year.
4. History of epilepsy, other neurological disorders, or neuropsychiatric conditions.
5. Subjects with ECG abnormalities (history, or evidence of second-degree heart block of Mobitz type II, third degree heart block, or any abnormality considered relevant by the Investigator), QTcF > 450 ms, PR > 210 ms, or QRS duration > 115 ms.
6. Supine systolic blood pressure > 140 mmHg or < 90 mmHg or diastolic blood pressure > 90 mmHg or < 50 mmHg at Screening or Day 1 prior to dosing (any abnormal blood pressure results may be repeated once and if the repeat result is within the normal range, it is not considered to have met the exclusion criterion). Pulse rate > 90 or < 50 beats per minute at Screening or Day 1 prior to dosing.
7. Glomerular Filtration Rate (GFR) < 80 mL/min/1.73m2 as calculated by the Chronic Kidney Disease Epidemiology Collaboration formula.
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and creatinine, above the upper limit of normal (ULN) at Screening. Any abnormal value of these parameters may be repeated and if the repeat result is within the laboratory reference range, it is not considered to have met the exclusion criterion.
9. Screening values other than AST, ALT, ALP, creatinine, for haematology, clinical chemistry, or urinalysis must not exceed the reference range. Minor deviations from normal are allowed, if they are not clinically significant.
10. History of symptomatic, chronic or recurrent infection (e.g. nausea, vomiting, diarrhoea, infection with fever) or any viral (including symptomatic herpes zoster), bacterial (including upper respiratory infection), fungal (non-cutaneous) or parasitic infection within 30 days prior to admission to the clinical unit.
11. Evidence of COVID-19 signs or symptoms, exposure to infected person or confirmed COVID-19 infection within the last 2 weeks.
12. Subjects who have received any prescribed systemic or topical medication within 4 weeks of the dose administration or within 5 times the half-life, whichever is longer, except for the occasional use of paracetamol (up to 2 g/day).
13. Subjects who have used any non-prescribed systemic or topical medication (including dietary supplements, natural and herbal remedies) or megadose vitamins (i.e. 20 to 600 times the recommended daily supplement dose) within 7 days of the dose administration, unless in the opinion of the Investigator the medication will not interfere with the trial procedures or compromise safety.
14. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration.
15. Regular use of any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to admission to the clinical unit.
16. Administration of live, attenuated, replication-competent vaccine(s), including vector-based or mRNA COVID-19 vaccine(s), within 1 month prior to screening or plans to receive such vaccines during the trial.
17. Subjects who have participated in a clinical trial involving administration of an investigational drug (new chemical entity) within the following time period prior to the dosing day in the current trial: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
18. Exposure to more than 4 new chemical entities in the last 12 months before the first dosing day in this trial.
19. A positive pre-study serology test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV)-1 and/or 2 antibodies.
20. A positive pre-study drug/alcohol screen/SARS-CoV-2 test. Higher than low-risk alcohol consumption i.e., consumption of an average weekly alcohol intake of 14 units/week for men (daily dose of 24 g, weekly dose of 168 g). One unit (12 g) corresponds to 0.3 L of beer/day or 0.12 L of wine/day or 1 glass (at 2 cL) of spirits/day.
21. Excessive consumption of caffeine- or xanthine-containing food or beverages (> 5 cups of coffee a day or equivalent) or inability to stop consuming from 48 hours prior to study treatment administration.
22. Any use of drugs-of-abuse or alcohol abuse within 2 years prior to the first admission to the clinical unit.
23. Subjects who are unable to refrain from the consumption of Seville oranges, grapefruit or grapefruit juice and /or pomelos, exotic citrus fruits, grapefruit hybrids, starfruit or fruit juices from 1 day prior to the first dose of Study Drug on Day 1, until completion of the last PK blood sample time point.
24. Inability to understand or communicate reliably with the Investigator or considered by the Investigator to be unable to or unlikely to co-operate with the requirements of the trial.
25. Any other conditions or factors which in the opinion of the Investigator may interfere with trial conduct. Failure to satisfy the Investigator of fitness to participate for any other reason.
26. Any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days prior to the first admission to the clinical unit.
27. Inability to refrain from using soft contact lenses starting from administration of study treatment until follow-up visit.
28. Subjects who are study site employees or immediate family members of the study site or Sponsor employee.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of increasing multiple intravenous doses of BV100 | 21 Days
  Incidence of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
To characterize the pharmacokinetic profile of rifabutin | 11 Days
  Area under the plasma concentration versus time curve (AUC)
To characterize the plasma concentration of rifabutin | 11 Days
  Peak Plasma Concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No